CLINICAL TRIAL: NCT01845194
Title: Open Label Repeated Dose Study for the Evaluation of Heritability of and Genetic Influences on Drug Pharmacokinetics (TWINS II)
Brief Title: Repeated Dose Study for the Investigation of Heritability of and Genetic Influences on Drug Pharmacokinetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institut fuer anwendungsorientierte Forschung und klinische Studien GmbH (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: TWINS-II-v1.9
Record Dates: First submitted 2013-04-25; First posted 2013-05-03 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Drug Biotransformation; Membrane Transport
Keywords: pharmacokinetic; heritability; drug membrane transport; drug biotransformation
MeSH Terms: interventions — Codeine; Midazolam; Pravastatin; Torsemide; talinolol; Caffeine; Metoprolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Drug application (Experimental): Two treatment periods:
  Treatment period 1:
  three sequential oral and i.v. doses of 5 mg Metoprolol, 50 mg Talinolol, 2.5 mg Torsemide, 0.2 mg Midazolam and 50 mg Caffeine. At least 1 week of wash out between drug application
  Treatment period 2:
  combined application of a single oral dose of 2.5 mg Talinolol, 0.25 mg Torsemide, 5 mg Pravastatin, 1 mg Midazolam and 5 mg Codeine.
  Treatment period 2 may take place after or before treatment period 1 with a time interval of at least 1 week
  Interventions: Drug: Codeine; Drug: Midazolam; Drug: Pravastatin; Drug: Torsemide; Drug: Talinolol; Drug: Caffeine; Drug: Metoprolol

INTERVENTIONS:
Drug: Codeine — Treatment period 2:
  5 mg Codeine once
Drug: Midazolam — Treatment period 1:
  0.2 mg Midazolam 3x
  Treatment period 2:
  1 mg Midazolam once
Drug: Pravastatin — Treatment period 2:
  5 mg Pravastatin once
Drug: Torsemide — Treatment period 1:
  2.5 mg Torsemide 3x
  Treatment period 2:
  0.25 mg Torsemide once
Drug: Talinolol — Treatment period 1:
  50 mg Talinolol 3x
  Treatment period 2:
  2.5 mg Talinolol once
Drug: Caffeine — Treatment period 1:
  50 mg Caffeine 3x
Drug: Metoprolol — Treatment period 1:
  5 mg Metoprolol 3x

SUMMARY:
This human pharmacokinetic study investigates, whether processes of drug metabolism and transport are determined by genetic or hereditary factors. Therefore, approved drugs are applied to twins and metabolism and transport processes are investigated.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained prior to study entry including informed consent for genetic research
* Both genders (male and female)
* Healthy adults aged ≥18 to < 65 years
* Body weight of subjects of both genders not less than 50 kg and not more than 120 kg. BMI not less than 18 kg/m² and not greater than 33 kg/m²
* Willingness to meet the study instructions and to co-operate with the study personal
* No clinically relevant pathological findings in any of the investigations at the Screening visit. Minor deviations of laboratory values from the normal range may be accepted, if judged by the investigator to have no clinical relevance
* Female subjects will only be included if they have negative serum pregnancy test during screening and the willingness not to become pregnant during the entire study period by practicing reliable methods of contraception as specified in the respective protocol section.
* Dizygotic twins will only be included if both siblings are of the same gender, either male or female and triplets, quadruplets or other multiplets if at least two siblings are of the same gender
* Smokers will only be included if both siblings are smoking to a similar extend (+/- 10 cigarettes per day)

Exclusion Criteria:

* Involvement in the planning and conduct of the study (applies to staff directly employed at the study site / department)
* Participation in a clinical study during the last 30 days or use of any other investigational or non-registered drug or vaccine during the study period or within 30 days preceding the first dose of study drugs
* Blood, plasma or thrombozyte donation during the last 30 days prior to application of the test drugs
* Age < 18 years or > 65 years
* Known pregnancy or lactation period
* Any relevant pathological findings in any of the investigations at the screening visit including significant abnormalities as result of the medical-screening-laboratory-analysis, especially of the liver and kidney related parameters.
* Any disease affecting liver or kidney or impairment of the liver or kidney-function
* Any cardiac disease in which use of beta-blockers or caffeine might be contraindicated.
* Bronchogenic asthma requiring constant drug treatment (stages 2 to 4 asthma)
* Known Raynaud's syndrome
* Any major acute disease or fever (Temp. > 37.5 C)
* Any major gastrointestinal disease and any gastrointestinal disorder that is expected to significantly interfere with the pharmacokinetics of the study drug
* Gastrointestinal surgery which may interfere with the pharmacokinetics of the study drug (except appendectomy or herniotomy)
* Taking any medication within 7 days before or during the trial with the following exceptions: Single doses of mild analgesics (e.g. aspirin, paracetamol, ibuprofen) may have been taken except for the time from 6 hours prior to taking the test drug until 24 hours after taking the test drug. Oral contraceptive drug used will be documented but will not be an exclusion criterion. Other medication might be allowed on single case basis if considered necessary for the subject's safety and well-being.
* History of alcohol and/or drug addiction and/or any abusive use of medicaments and/or positive drug screen
* Any other findings that could compromise the safety of the participant or the quality of the study-results
* History of severe hypersensitivity reactions and anaphylaxis
* If hypersensitivity or allergic reactions to one of the IMPs is known so enrolment is possible but application of the concerned IMP must not be allowed in all siblings (e.g. allergy to sulphonamide prohibits specifically the application of torsemide)
* Clinically significant diseases as judged by the investigator
* Body temperature > 37.5°C prior to drug application
* Known infection with HIV, Hepatitis B (HBsAg) or Hepatitis C
* Inability or unwillingness to avoid any intake of alcohol from 48h prior to until 72hours after IMP application
* Pregnancy (positive pregnancy test during screening and/or treatment)
* Lactation or unreliable contraception in female subjects with child-bearing potential
* Inability or unwillingness to provide informed consent and to abide by the requirements of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2009-12; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
plasma drug concentrations | up to 24 h after drug application
  Up to 8 (± 60 min.) hour after each application of combined drugs (treatment period 1 and treatment period 2) blood and urine collection is continuously performed and drug concentrations as specified in the sections "study arms" and "interventions" are measured. This is repeated once 24 hours after each drug application.

SECONDARY OUTCOMES:
PK and metabolic ratios | up to 24 h after drug application
  PK and metabolic ratios (MR, ratio between parent compound and metabolite) of the test substrates as specified in the sections "study arms" and "interventions" are measured.
variants in known genetic traits | up to 24 h after drug application
  New variants in known genetic traits are investigated and new genetic traits are identified.
design applicability | 54 months after study start
  To evaluate the applicability of the repeated measure design for other, non drug-related genetic traits, such as blood coagulation pathways.

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Brockmöller, Prof., Study Chair — Dept. of Clinical Pharmacology, Georg-August-University of Goettingen, Robert-Koch-Str. 40, 37075 Goettingen, Germany
Locations (1):
- Dept. of Clinical Pharmacology, Georg-August-University of Goettingen, Göttingen, Germany

REFERENCES:
- [Derived] Matthaei J, Bonat WH, Kerb R, Tzvetkov MV, Strube J, Brunke S, Sachse-Seeboth C, Sehrt D, Hofmann U, von Bornemann Hjelmborg J, Schwab M, Brockmoller J. Inherited and Acquired Determinants of Hepatic CYP3A Activity in Humans. Front Genet. 2020 Aug 21;11:944. doi: 10.3389/fgene.2020.00944. eCollection 2020. PMID 32973880
- [Derived] Matthaei J, Tzvetkov MV, Gal V, Sachse-Seeboth C, Sehrt D, Hjelmborg JB, Hofmann U, Schwab M, Kerb R, Brockmoller J. Low heritability in pharmacokinetics of talinolol: a pharmacogenetic twin study on the heritability of the pharmacokinetics of talinolol, a putative probe drug of MDR1 and other membrane transporters. Genome Med. 2016 Nov 8;8(1):119. doi: 10.1186/s13073-016-0372-2. PMID 27825374
- [Derived] Matthaei J, Brockmoller J, Tzvetkov MV, Sehrt D, Sachse-Seeboth C, Hjelmborg JB, Moller S, Halekoh U, Hofmann U, Schwab M, Kerb R. Heritability of metoprolol and torsemide pharmacokinetics. Clin Pharmacol Ther. 2015 Dec;98(6):611-21. doi: 10.1002/cpt.258. Epub 2015 Oct 19. PMID 26344676